CLINICAL TRIAL: NCT00525850
Title: Effect of High Saturated Fat No Starch Diet vs. Low Saturated Fat, Low Trans Fat, High Fiber Diet on Weight Loss and Markers of Atherosclerotic Cardiovascular Disease
Brief Title: High Fat Diet II on Weight Loss
Acronym: HFD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Angela DiSabatino, RN, MS, Manager, Cardiovascular Clinical Trials Program, Christiana Care Health Services
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCC26177
Record Dates: First submitted 2007-09-05; First posted 2007-09-06 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-08

CONDITIONS: Obesity
Keywords: cardiovascular disease; weight loss
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Weight Loss | interventions — Diet, High-Fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): high saturated fat diet
  Interventions: Other: high fat diet
- 2 (Other): low calorie low saturated fat low trans fat high fiber diet
  Interventions: Other: low saturated fat diet

INTERVENTIONS:
Other: high fat diet — high saturated fat no starch diet
  Arms: 1
Other: low saturated fat diet — low calorie low saturated fat low trans fat high fiber diet
  Arms: 2

SUMMARY:
To evaluate two different diets and their effects on weight loss and measurements of several risk factors for cardiovascular disease. One diet will be a high saturated fat diet (HSFD) and the other is a low saturated fat diet (LSFD) that limits fat but especially saturated fat as red meat. All participants in this study must eat both diets as this is a randomized cross-over design.

ELIGIBILITY:
Inclusion Criteria:

In order to qualify, participants must have metabolic syndrome:

* triglycerides greater than 150 mg/dL
* blood pressure greater than 130 mmHg and/or diastolic blood pressure greater than 85 mmHg
* fasting glucose greater than 110 mg/dL
* waist circumference greater than 40 inches in men or 35 inches in women
* reduced HDL less than 40 mg/dL in men and less than 50 mg/dL in women. Participants must be capable of performing symptom-limited maximal exercise capacity study. Blood and urine samples collected at baseline will be analyzed for CBC, serum glucose and electrolytes, hepatic panel and TSH.

Exclusion Criteria:

Participants will be excluded for any significant blood dyscrasia, fasting glucose greater than 200 mg/dL, creatine greater than 2 mg/dL, any significant electrolyte disorder, hepatic functions greater than two times normal or abnormal TSH.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Weight loss | 12 weeks

SECONDARY OUTCOMES:
Brachial artery reactivity | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James Hays, MD, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care Health System, Newark, Delaware, United States